CLINICAL TRIAL: NCT03951441
Title: Construct Validity and Reliability of the Selective Control Assessment of the Lower Extremity in Children With Cerebral Palsy
Brief Title: Construct Validity and Reliability SCALE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve TUNÇDEMİR, Research Assisstant, Hacettepe University
Other Study IDs: selectivemotorcontrol
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Palsy
Keywords: lower limb
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to determine construct validity, discriminant validity and intra- and interrater reliability of the Selective Control Assessment of the Lower Extremity ( SCALE).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of spastic cerebral palsy,
* age between 4 and 18 years,
* ability to follow simple instructions.
* ability to walk (GMFCS levels I-IV),

Exclusion Criteria:

* unstable situation regarding their tonus-regulating medications
* orthopedic intervention or surgical correction within the last year,
* botulinum toxin injection within the last 6 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Spastic Cerebral Palsy
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-06-20 (Estimated); Study Completion 2019-07-22 (Estimated)

PRIMARY OUTCOMES:
Selective Control Assessment of the Lower Extremity | 15 minutes
  SCALE examines SVMC in children with spastic CP. The SCALE tool assesses hip, knee, ankle, subtalar, and toe joints bilaterally.The SCALE tool assigns each joint a score from 0 to 2 points: 2 points, normal; 1 point, impaired; and 0 points, unable. The SCALE score is the sum of scoresfor each joint and assumes a 10 point maximum per limb.

SECONDARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | 2 minutes
  The GMFCS describes gross motor function in children with CP. It focuses on self-initiated movements, in particular sitting and walking. It is an age-related five-level system in which level I represents the least limitation and level V the most.
Gross Motor Function Measurement (GMFM) | 15 minutes
  Gross Motor Function Measurement evaluates motor functions in children with Cerebral Palsy. There is 88 items under 5 subdimensions (lying and rolling, sitting, crawling and kneeling, standing, walking-running-jumping. GMFM has a 4-point scoring system for each item. The higher the child gets, the more successful the child is in gross motor functions.
Modified Ashworth Scale (MAS) | 5 minutes
  Tone of lower extremity muscles will be assessed with Modified Ashworth Scale. The spasticity of each muscle ranged between 0 to 5. 0 means no increase in muscle tonus while 5 means that the joint is rigid due to the increase in excess tonus.
The Physicians' Rating Scale (PRS) | 5 minutes
  The Physicians' Rating Scale is an observational tool that has been used to evaluate gait. PRS is assesses gait in the sagittal plane.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)